CLINICAL TRIAL: NCT05194254
Title: MRI-Eye Tracking Pairing, a Tool for Assessing Social Cognition in Children With ASD
Acronym: IRM-ET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2021_843_0194
Record Dates: First submitted 2022-01-04; First posted 2022-01-18 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: ASD; Functional Magnetic Resonance Imaging; Eye Tracking; Social Cognition; Joint Attention
Keywords: ASD; Functional magnetic resonance imaging; Eye Tracking; social cognition; joint attention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ASD (Experimental): people with Autism Spectrum Disorders
  Interventions: Other: MRI-ET
- TD (Active Comparator): Typical Development) group of people
  Interventions: Other: MRI-ET

INTERVENTIONS:
Other: MRI-ET — coupled fMRI and Eye Tracking tools

SUMMARY:
Most studies use static visual percepts that are less representative of joint attention versus an ecological environment. This has the consequence of decreasing the perception of an interaction with a social partner, which is an essential step in achieving joint attention. The originality of this study is to improve the design of visual percepts (in the form of video) in order to mimic an ecological environment as much as possible by using MRI-ET coupling. The second originality of this study is the longitudinal exploration of the neurodevelopment of social cognition in autistic children. Studies by the Redcay and Oberwelland teams observe different activations at different ages. The hypothesis is that the perception of joint attention varies over time in people with ASD. To date, there are no studies to determine the influence of childhood neurodevelopment in autistic people on the perception of joint attention. It would be unprecedented to use the MRI-ET pairing as a tool for assessing social cognition as a function of the development of children with ASD.

ELIGIBILITY:
Inclusion Criteria:

For the group of people with Autism Spectrum Disorders (experimental group):

* Age between 10 to 20 years old
* Diagnosis of ASD (CARS) ≥ 30 performed at inclusion
* IQ test evaluation (regardless of the result) performed by a trained psychologist
* Obtaining informed oral and written consent after appropriate information
* Obtaining informed oral and written consent from the legal guardian after information
* Be affiliated with social security
* No contraindication to magnetic resonance imaging

For the TD (Typical Development) group of people (control group):

* Age between 10 to 20 years old
* Diagnosis of ASD (CARS) <30 performed at inclusion
* IQ test evaluation (regardless of the result) performed by a trained psychologist
* Obtaining informed oral and written consent after appropriate information
* Obtaining informed oral and written consent from the legal guardian after information
* Be affiliated with social security
* No contraindication to magnetic resonance imaging

Exclusion Criteria:

For all groups:

* Age outside the range 10 to 20 years
* Person with a contraindication to MRI (including claustrophobia, pace maker, neurosurgical clips, vascular clips, heart valves, ventriculoperitoneal valves, cochlear implant, neurostimulator, intraocular metal shards, joint prosthesis, etc.)
* Person suffering from major obesity (> 140 kg) not allowing him to enter the tunnel of the MRI machine (diameter <70cm)
* Pregnant or breastfeeding woman
* Person under guardianship or guardianship or deprived of liberty by a judicial or administrative decision

For TD people (control group):

* Person with psychiatric disorders such as attention disorder with or without hyperactivity, depression, bipolar disorder and schizophrenia.
* Person with a neurological history such as epilepsy and / or neurovascular accident.

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-01-04 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
difference of mapping IRM-ET results between both patient groups | one day
  both patient groups are : the group of people with Autism Spectrum Disorders and Typical Development group of people

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No